CLINICAL TRIAL: NCT02840253
Title: Changes in Tissue and Cerebral Oxygenation Following Spinal Anesthesia in Neonates, Infants, and Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joseph D. Tobias (Other)
Responsible Party: Sponsor-Investigator, Joseph D. Tobias, Chairman, Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB16-00465
Record Dates: First submitted 2016-06-23; First posted 2016-07-21 (Estimated); Results first posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Infants Undergoing Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NIRS (Experimental): Non-invasive near infrared spectroscopy to assess changes in tissue and cerebral oxygenation.
  Interventions: Device: NIRS

INTERVENTIONS:
Device: NIRS

SUMMARY:
Investigators have started an awake spinal anesthesia program in conjunction with pediatric surgical colleagues. Patients are offered the option of awake spinal anesthesia instead of general anesthesia for appropriate surgical procedures. Previous studies have demonstrated a lack of significant hemodynamic changes in neonates and infants following spinal anesthesia; however, there are limited data regarding its impact on tissue oxygenation. The goal of the current study is to assess changes in tissue and cerebral oxygenation using non-invasive near infrared spectroscopy following spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* All patients that are candidates for and have agreed to spinal anesthesia.

Exclusion Criteria:

* none

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-05-12 (Actual); Study Completion 2017-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Tobias, MD, Principal Investigator — Nationwide Children's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Froyshteter AB, Tumin D, Whitaker EE, Martin DP, Hakim M, Walia H, Bhalla T, Tobias JD. Changes in tissue and cerebral oxygenation following spinal anesthesia in infants: a prospective study. J Anesth. 2018 Apr;32(2):288-292. doi: 10.1007/s00540-017-2446-8. Epub 2018 Jan 12. PMID 29330639

RESULTS

PARTICIPANT FLOW:
Groups:
- NIRS: Non-invasive near infrared spectroscopy to assess changes in tissue and cerebral oxygenation.
  NIRS
Period: Overall Study
Arm/Group | NIRS
Started | 23
Completed | 19
Not Completed | 4
Not completed — Unsuccessful block | 4

BASELINE CHARACTERISTICS:
Population: 4 subjects had unsuccessful blocks
Arm/Group | NIRS
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: months] | 7 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Cerebral Non-invasive Near Infrared Spectroscopy (NIRS)
Description: Change in cerebral oxygen saturation from immediately after spinal anesthesia placement to conclusion of monitoring (30 mins post block).
Time Frame: Intraoperative measure
Measure: Number (95% Confidence Interval); unit: percentage change per minute
Arm/Group | NIRS
Number analyzed (Participants) | 19
percentage change per minute | 0.05 [-0.1 to 0.19]

2. Primary Outcome: Tissue Non-invasive Near Infrared Spectroscopy (NIRS)
Description: Change in tissue oxygen saturation from immediately after spinal anesthesia placement to conclusion of monitoring (30 mins post block).
Time Frame: Intraoperative measure
Measure: Number (95% Confidence Interval); unit: percentage change per minute
Arm/Group | NIRS
Number analyzed (Participants) | 19
percentage change per minute | 0.04 [0.01 to 0.08]

ADVERSE EVENTS:
Time Frame: Until discharge to home, approximately 2 hours.
Arm/Group | NIRS
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-14): https://cdn.clinicaltrials.gov/large-docs/53/NCT02840253/Prot_SAP_000.pdf